CLINICAL TRIAL: NCT04341896
Title: The Role of Caregiving in Healthcare Utilization Among Obese Living Kidney Donors
Brief Title: Healthcare Utilization in Obese Caregiver Living Donors
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rhiannon Deierhoi Reed, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300000039; P30AG031054 (NIH)
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Utilization, Health Care; Obesity
Keywords: living kidney donor
MeSH Terms: conditions — Patient Acceptance of Health Care; Obesity | interventions — Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caregivers: Prior obese living kidney donors who served as the primary caregiver for their recipient
  Interventions: Other: Caregivers
- Non-caregivers: Prior obese living kidney donors who were not the primary caregiver for their recipient
  Interventions: Other: Non-caregivers

INTERVENTIONS:
Other: Caregivers — Individuals who cared for themselves and their transplant recipient before and after kidney donation
  Groups: Caregivers
Other: Non-caregivers — Individuals who donated a kidney as a living donor but did not serve as the primary caregiver for their recipient
  Groups: Non-caregivers

SUMMARY:
The goal of this study is to estimate risk of post-donation healthcare use attributable to informal caregiving among obese living donors. Improving our understanding of the relationship between caregiving, donation, and healthcare use will allow us to improve living donor informed consent and post-donation care, particularly among older donors and those of minority race/ethnicity.

DETAILED DESCRIPTION:
Caregiver burden is a well-known issue of primary caregiving for individuals with chronic disease, including transplant candidates and recipients. Informal caregiving is associated with an estimated $306 billion in unpaid labor costs and an average of $7,000 in out-of-pocket expenses related to the caregiving role. In addition to financial burdens, caregivers experience psychological distress and adverse health outcomes, including higher rates of hypertension and heart disease. These burdens differ by caregiver ethnicity, age, and rurality. Ethnic minority caregivers have reported more depression, lower use of support services, and worse physical health than Whites. African American caregivers report lower levels of depression but worse physical health. Caregiver age also plays a role in physical health burden, with older caregiver age shown to be negatively associated with caregiver physical functioning, bodily pain, vitality, and general health perception. This association is directly relevant to living kidney donation, as the prevalence of donors who are 65 years or older has increased from < 1% in 1998 to 5.6% in 2019 (based on OPTN data as of 3/23/2020). Rural caregivers report greater financial burden than their urban counterparts, of particular concern in the Deep South, where nearly two-thirds of all counties are rural.

When caregivers have their own underlying health issues, such as obesity, burdens may be further magnified when the caregiver becomes a patient, simultaneously requiring their own care while caring for another (e.g. obese living kidney donors who are the primary caregiver for their transplant recipient). Approximately 20% of living kidney donors are parents and significant others, individuals who often serve as the recipient's primary caregiver. Moreover, obese donors are at higher risk of post-donation disease development, including end-stage renal disease, diabetes, and hypertension. As donor selection criteria have expanded to include more obese individuals, these burdens impact high volume transplant centers in the Deep South that serve largely minority and rural populations. Comorbidity, such as obesity, in caregiver donors may increase the need for healthcare utilization, further exacerbating financial burdens, interfering with caregiver responsibilities, and subsequently impacting the recipient's health outcomes. To date, it is unknown whether the burdens of being an obese caregiver living donor are associated with healthcare utilization post-donation compared to non-caregivers and whether donor age, race, and rurality modify this relationship. This study is ancillary to an NIH-funded retrospective cohort study of living kidney donors with obesity (1R01DK113980) and will leverage the infrastructure of this R01 to explore the primary exposure of caregiving within this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Underwent living donor nephrectomy at a transplant center in the United States between 1968 to present
* Obesity: had a body mass index of 30 kg/m2 or greater at time of kidney donation

Exclusion Criteria:

* Age < 18 years
* Non-obese at time of donation
* Does not consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is an ancillary study to 1R01DK113980, a retrospective cohort study that is assembling the largest cohort of previous living kidney donors with obesity from 1968-present from all centers across the US. The parent R01 is projected to enroll approximately 25,000 obese living donors, and 20% (n=5,070) of these are estimated to have served as the primary caregiver for their transplant recipient (the primary exposure of this study).
Sampling Method: Non-Probability Sample
Enrollment: 784 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhiannon Reed, DrPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caregivers | Non-caregivers
Started | 148 | 636
Completed | 148 | 636
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: These numbers correspond to the individuals who completed survey measures during the study period and indicated whether or not they were the primary caregiver for their transplant recipient.
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregivers | Non-caregivers | Total
Number analyzed (Participants) | 148 | 636 | 784
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 49.1 [42.8 to 55.7] | 46.5 [38.2 to 54.3] | 47.2 [39.1 to 54.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 371 | 474
  Male | 45 | 265 | 310
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 3 | 10 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 64 | 80
  White | 124 | 529 | 653
  More than one race | 3 | 27 | 30
  Unknown or Not Reported | 1 | 2 | 3
Relationship to recipient [Count of Participants; unit: Participants]
  Parent | 24 | 29 | 53
  Spouse/partner | 74 | 50 | 124
  Child | 14 | 76 | 90
  Sibling | 19 | 163 | 182
  Other biologic | 3 | 69 | 72
  Non-biologic | 14 | 249 | 263
Working for income [Count of Participants; unit: Participants]
  Part-time | 11 | 50 | 61
  Full-time | 66 | 383 | 449
  Unemployed | 13 | 43 | 56
  Retired | 56 | 158 | 214
  Unknown | 2 | 2 | 4
Marital status [Count of Participants; unit: Participants]
  Single | 31 | 101 | 132
  Married | 86 | 435 | 521
  Co-habitating | 6 | 20 | 26
  Divorced | 14 | 66 | 80
  Unknown | 11 | 14 | 25
Time since donation [Median (Inter-Quartile Range); unit: Years] | 11.8 [5.8 to 17.1] | 10.3 [5.8 to 15.1] | 10.4 [5.8 to 15.4]

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department Utilization
Description: Proportion self-reporting at least one visit to the emergency department since donation/previous questionnaire
Time Frame: 44 months
Population: The denominator for this outcome is based on participants who responded to the survey item asking about emergency department utilization since donation
Measure: Count of Participants; unit: Participants
Arm/Group | Caregivers | Non-caregivers
Number analyzed (Participants) | 144 | 618
Participants | 77 | 305

2. Primary Outcome: Hospital Admission
Description: Proportion self-reporting at least one hospital admission since donation/previous questionnaire
Time Frame: 44 months
Population: The denominator is from participants who responded to the survey question regarding hospitalization since donation.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregivers | Non-caregivers
Number analyzed (Participants) | 138 | 588
Participants | 71 | 237

ADVERSE EVENTS:
Time Frame: 44 months
Description: This was a retrospective survey, and as such, the only potential risk was accidental breach of confidentiality. No adverse events occurred.
Arm/Group | Caregivers | Non-caregivers
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/636
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/636
Other Adverse Events (participants affected / at risk) | 0/148 | 0/636

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT04341896/Prot_SAP_000.pdf